CLINICAL TRIAL: NCT00004921
Title: A Randomized Phase III Trial of Sequential High Dose Chemotherapy or Standard Chemotherapy for Optimally Debulked FIGO Stage III and IV Ovarian Cancer
Brief Title: High-Dose Chemotherapy Compared With Standard Chemotherapy in Treating Patients With Stage III or Stage IV Ovarian Epithelial Cancer That Has Been Removed During Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EBMT Solid Tumors Working Party (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067604; EBMT-HIDOC-EIS; EBMT-OVCAT; EU-99040
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2002-07

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Melphalan; Paclitaxel; Chemotherapy, Adjuvant; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: melphalan
Drug: paclitaxel
Procedure: adjuvant therapy
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is most effective for ovarian epithelial cancer.

PURPOSE: This randomized phase III trial is studying high-dose chemotherapy to see how well it works compared to standard chemotherapy in treating patients with stage III or stage IV ovarian epithelial cancer that has been removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the two-year progression-free survival in patients with optimally debulked stage III or IV ovarian epithelial cancer undergoing high-dose sequential chemotherapy vs standard chemotherapy.
* Compare the overall survival, toxicity, and quality of life in this patient population receiving these two treatment regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive 5 courses of sequential high-dose chemotherapy as follows:

  * Courses 1 and 2: Patients receive paclitaxel IV over 3 hours and cyclophosphamide IV over 2 hours on day 1 followed by peripheral blood stem cell (PBSC) collection. Patients receive filgrastim (G-CSF) subcutaneously (SC) beginning 24 hours following chemotherapy and continuing until target number of PBSC are reached.
  * Courses 3 and 4: Patients receive paclitaxel as in courses 1-2 and carboplatin IV over 4 hours on day 1. At 72 hours following completion of carboplatin, patients receive PBSC infusion. Beginning one day following PBSC infusion, patients receive G-CSF SC until blood counts recover.
  * Course 5: Patients receive paclitaxel as in courses 1 and 2 and carboplatin as in courses 3 and 4 and melphalan IV over 15 minutes on day 2 or 3. Patients receive PBSC and G-CSF as in courses 3 and 4.
  * Treatment repeats every 3-4 weeks.
* Arm II: Patients receive standard chemotherapy consisting of carboplatin (or cisplatin) and paclitaxel IV over 3 hours every 3 weeks for 6 courses. Patients may receive doxorubicin or epirubicin in addition to the standard chemotherapy every 4 weeks.

Quality of life is assessed prior to therapy, at 4-6 weeks following completion of therapy, and then at 3 months, 9 months, and 15 months.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 208 patients (104 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV ovarian epithelial cancer
* Bilateral salpingo-oophorectomy, hysterectomy, and omentectomy within 6 weeks of study

  * Less than 2 cm maximum diameter of residual tumor remaining

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Normal hematological function

Hepatic:

* Normal hepatic function

Renal:

* Creatinine clearance greater than 60 mL/min
* GFR greater than 60 mL/min

Cardiovascular:

* No active cardiac disease

Other:

* No other uncontrolled serious medical illness, including hearing problems
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A. Ledermann, MD, Study Chair — Cancer Research UK
Locations (17):
- Sozialmedizinisches Zentrum Ost - Donauspital, Vienna, Austria
- Centre Hospitalier Notre Dame - Reine Fabiola, Charleroi, Belgium
- Czechia (2):
  - Charles University, Prague
  - Thomayer Memorial Teaching Hospital, Prague
- Germany (2):
  - Staedt Klinikum Karlsruhe GGMBH, Karlsruhe
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
- Italy (4):
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Ospedale Santa Chiara, Pisa
  - S. Camillo Hospital, Rome
  - Ospedale San Bortolo, Vicenza
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Spain (2):
  - Hospital Universitario San Carlos, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (3):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Cancer Research UK and University College London Cancer Trials Centre, London, England
  - Cancer Research Centre at Weston Park Hospital, Manchester, England

REFERENCES:
- [Result] Mobus V, Wandt H, Frickhofen N, Bengala C, Champion K, Kimmig R, Ostermann H, Hinke A, Ledermann JA; AGO-Ovar/AIO; EBMT. Phase III trial of high-dose sequential chemotherapy with peripheral blood stem cell support compared with standard dose chemotherapy for first-line treatment of advanced ovarian cancer: intergroup trial of the AGO-Ovar/AIO and EBMT. J Clin Oncol. 2007 Sep 20;25(27):4187-93. doi: 10.1200/JCO.2006.09.7527. Epub 2007 Aug 13. PMID 17698804